CLINICAL TRIAL: NCT00362596
Title: A Randomized Controlled Crossover Trial of Acylcovir Among HIV and HSV-2 Co-Infected Women, Chiang Rai, Thailand
Brief Title: A Randomized Controlled Trial of Acyclovir Among HIV and HSV-2 Co-Infected Women, Chiang Rai, Thailand
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health, Thailand (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-4178
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Last update posted 2006-08-10 (Estimated); Status verified 2006-08

CONDITIONS: HIV; Herpes
Keywords: Acyclovir; HIV; HSV
MeSH Terms: conditions — Herpes Simplex | interventions — Acyclovir

INTERVENTIONS:
Drug: acyclovir

SUMMARY:
Herpes infection is an important co-factor in HIV transmission. A recent meta-analysis demonstrated that HSV infection contributed to a 2-fold increased risk of HIV transmission. Suppressive therapy with acyclovir has been a method proposed to reduce HIV transmission. We are conducting a randomized controlled cross-over trial to evaluate the effect of acyclovir suppressive therapy on HIV genital shedding in women co-infected with HIV-1 and Herpes Simplex Virus Type-2 (HSV-2) in Thailand.

DETAILED DESCRIPTION:
65 women ages 18-49 years old with HIV-1 and HSV-2 co-infection are being recruited from general medicine clinics, family planning clinics, postnatal clinics, community based organizations and community outreach in Chiang Rai, Thailand.

Our study objectives are:

* To evaluate the effect of acyclovir suppressive therapy on HIV genital shedding.
* To determine the association between HIV and HSV genital shedding, and the effect of acyclovir suppressive therapy on this association.
* To determine the acceptability of acyclovir suppressive therapy for women with HIV infection.
* To evaluate the association of genital symptoms and HIV or HSV genital shedding.
* To evaluate the association between cervicovaginal (CVL) specimens and self-collected genital swabs for detection of HIV and HSV-2.

ELIGIBILITY:
Inclusion Criteria:

* participants will be HIV and HSV-2 seropositive

Exclusion Criteria:

* pregnancy, CD4 count <200, on ART

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67
Dates: Start 2005-01; Study Completion 2005-08

PRIMARY OUTCOMES:
To evaluate the effect of acyclovir suppressive therapy on HIV genital shedding.

SECONDARY OUTCOMES:
To determine the association between HIV and HSV genital shedding, and the effect of acyclovir suppressive therapy on this association.
To determine the acceptability of acyclovir suppressive therapy for women with HIV infection.
To evaluate the association of genital symptoms and HIV or HSV genital shedding.
To evaluate the association between cervicovaginal (CVL) specimens and self-collected genital swabs for detection of HIV and HSV-2.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen F. Dunne, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention; Sara Whitehead, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- TUC, Chiang Rai, Changwat Chiang Rai, Thailand

REFERENCES:
- [Derived] Dunne EF, Whitehead S, Sternberg M, Thepamnuay S, Leelawiwat W, McNicholl JM, Sumanapun S, Tappero JW, Siriprapasiri T, Markowitz L. Suppressive acyclovir therapy reduces HIV cervicovaginal shedding in HIV- and HSV-2-infected women, Chiang Rai, Thailand. J Acquir Immune Defic Syndr. 2008 Sep 1;49(1):77-83. doi: 10.1097/QAI.0b013e3181831832. PMID 18667923